CLINICAL TRIAL: NCT03757312
Title: A Pilot Study of Optic Nerve Ultrasound Following Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marco Corridore (Other)
Responsible Party: Sponsor-Investigator, Marco Corridore, Associate Professor of Anesthesiology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB18-01209
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Results first posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Congenital Heart Disease; Congenital Heart Defect
Keywords: cardiopulmonary bypass
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fontan (Experimental): Patients undergoing Fontan procedure to redirect blood flow from the lower body to the lungs.
  Interventions: Diagnostic Test: Ultrasound
- Non-Fontan (Active Comparator): Patients undergoing other cardiac surgeries requiring cardiopulmonary bypass.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Ocular ultrasound to measure optic nerve sheath diameter (ONSD).

SUMMARY:
The purpose of the proposed study is to evaluate the incidence of subtle increases in intracranial pressure (ICP) following cardiopulmonary bypass (CPB) using optic nerve sheath diameter (ONSD), measured by non-invasive ultrasound. As direct measurements of ICP are not feasible following CPB, ONSD will be used as a correlate of ICP. ONSD has been shown to be effective in the ICU and emergency room setting for detecting increased ICP and is an accepted standard for such measurements. The primary hypothesis is that changes in ICP occur following CPB without clinically appreciable signs and symptoms. These changes in ICP will be reflected by changes in ONSD. If there is a significant incidence of sub-clinical cerebral edema and increased ICP postoperatively, these findings may impact postoperative hemodynamic and ventilation goals and techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 18 years of age undergoing cardiac bypass.

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Corridore, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fontan | Non-Fontan
Started | 5 | 9
Completed | 5 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fontan | Non-Fontan | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 9 | 14
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 2.6 [1 to 3] | 1.3 [0 to 6] | 1.8 [0 to 6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 2 | 5 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 9 | 14
Weight [Mean (Full Range); unit: kilograms] | 13.5 [7.9 to 16.6] | 9.3 [3.7 to 20.2] | 10.8 [3.7 to 20.2]
Height [Mean (Full Range); unit: centimeters] | 88.2 [63 to 97.1] | 74.3 [53 to 114.6] | 79.2 [53 to 114.6]
American Society of Anesthesiologists (ASA) status [Count of Participants; unit: Participants] — ASA 1 - normal healthy patient, ASA 2 - mild disease, ASA 3 - severe systemic disease, ASA 4 - severe systemic disease that is a constant threat to life
  Participants
    ASA 3 | 0 | 2 | 2
    ASA 4 | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Optic Nerve Sheath Diameter
Description: Optic nerve sheath diameter normal values: ≤4.0 mm for patients <1 year and ≤4.5 mm used for patients ≥1 year of age, thus there is potential for worse outcomes with higher diameters.
Time Frame: Day of surgery
Measure: Mean (Full Range); unit: millimeters
Arm/Group | Fontan | Non-Fontan
Number analyzed (Participants) | 5 | 9
millimeters
  Post induction of anesthesia | 4.0 [3 to 4.6] | 3.6 [3.1 to 3.9]
  After coming off of CPB | 4.2 [3.5 to 5.1] | 3.5 [3.1 to 3.9]
  Following tracheal extubation in the OR | 4.2 [3.2 to 5.3] | 3.7 [3.0 to 4.3]

2. Secondary Outcome: Optic Nerve Sheath Diameter: Short Versus Long Cardiopulmonary Bypass (CPB) Time
Description: Short CPB time defined as <100 minutes. Long CPB time defined as ≥ 100 minutes.
Time Frame: Day of surgery
Measure: Mean (Full Range); unit: millimeters
Groups:
- Short CPB Time: Short CPB time defined as <100 minutes.
- Long CPB Time: Long CPB time defined as ≥ 100 minutes.
Arm/Group | Short CPB Time | Long CPB Time
Number analyzed (Participants) | 7 | 7
millimeters
  Post-induction of anesthesia | 3.8 [3.6 to 4.0] | 3.6 [3.0 to 4.6]
  After coming off of CPB | 3.6 [3.5 to 3.9] | 3.8 [3.1 to 5.1]
  Following tracheal extubation in the OR | 3.8 [3.5 to 4.3] | 3.8 [3.0 to 5.3]

ADVERSE EVENTS:
Time Frame: 24 hours post-op
Arm/Group | Fontan | Non-Fontan
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 0/5 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT03757312/Prot_SAP_000.pdf